CLINICAL TRIAL: NCT01360203
Title: Variations in Care: Comparing Heart Failure Care Transition Intervention Effects
Brief Title: Better Effectiveness After Transition - Heart Failure
Acronym: BEAT-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Cedars-Sinai Medical Center (Other); University of California, Davis (Other); University of California, Irvine (Other); University of California, San Diego (Other); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Michael Ong, Associate Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R01HS019311 (AHRQ)
Record Dates: First submitted 2011-05-18; First posted 2011-05-25 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2014-05

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Remote Patient Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Current Care (No Intervention): Patients will receive the current care provided to heart failure patients at each of the study sites
- Care Transition Intervention (Experimental): Care transition intervention beginning prior to discharge and through six months post-discharge.
  Interventions: Other: Structured Telephone / Remote Outpatient Monitoring

INTERVENTIONS:
Other: Structured Telephone / Remote Outpatient Monitoring — During their hospitalization, patients will receive education on their condition and will be taught to use a wireless remote monitoring device that they will use from home on a daily basis for six months following hospital discharge. Patients will receive structured telephone phone calls from a centralized call center nurse at least once a week for the first month post-discharge, and monthly for the remainder of the six month study period. Patients may receive additional calls depending upon the information gathered during the scheduled call center phone calls and/or their health status as ascertained by the data (weight, heart rate, blood pressure, answers to general health and heart failure-related questions) transmitted daily by the wireless remote monitoring device.
  Other Names: Care Transition Intervention; Care Transitions Intervention; Structured Telephone Monitoring; Remote Monitoring
  Arms: Care Transition Intervention

SUMMARY:
The purpose of this study is to compare the effect of implementing wireless remote monitoring combined with structured telephone monitoring, versus current care, on variation in rehospitalization among older patients hospitalized with heart failure at six medical centers.

ELIGIBILITY:
Inclusion Criteria:

* patients hospitalized at any of the six medical centers who are being actively treated for heart failure.

Exclusion Criteria:

* patients who have previously received a transplant, are being evaluated for a transplant, or who are on the wait list for a transplant,
* patients who are enrolled or enrolling in hospice, or are expected to expire shortly after discharge,
* patients with dementia,
* patients who are admitted from a skilled nursing facility (SNF), or who we anticipate will be discharged to a long term stay in a SNF,
* patients who do not have a working land line phone or reliable cell service,
* patients on chronic dialysis,
* patients who cannot identify a usual source of care (free clinic is acceptable) and who will not be assigned a provider upon discharge,
* patients with the following cardiovascular conditions: patients with valvular disorders requiring surgical intervention (except for those with incidental valvular disease, who will be included), acute myocardial infarction (except for those with demand ischemia, who will be included), percutaneous coronary intervention
* patients expected to enroll in hospice or expire after discharge,
* patients who are unable to use the intervention equipment (e.g., unable to stand on the weight scale), or who are otherwise unable to comply with the intervention

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1437 (Actual)
Dates: Start 2011-10; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
180 day rehospitalization rate | at 180 days post-discharge
  Patient self-report in response to telephone survey, combined with administrative claims data of rehospitalization for any cause

SECONDARY OUTCOMES:
7 day mortality rate | within 7 days post-discharge
  Mortality during the study period. Next of kin will be contacted in the event the patient has expired to verify death and date of death.
Change in quality of Life | as an inpatient, within 7 days post-discharge, and at 30 and 180 days post-discharge
  Quality of life scores will be measured using standardized questionnaires, and data captured during enrollment will be compared with data captured during three post-discharge phone calls
30 day mortality rate | at 30 days post-discharge
  Mortality during the study period. Next of kin will be contacted in the event the patient has expired to verify death and date of death.
180 day mortality rate | at 180 days post-discharge
  Mortality during the study period. Next of kin will be contacted in the event the patient has expired to verify death and date of death.
30 day rehospitalization rate | at 30 days post-discharge
  Patient self-report in response to telephone survey, combined with administrative claims data of rehospitalization for any cause
7 day rehospitalization rate | within 7 days post-discharge
  Patient self-report in response to telephone survey, combined with administrative claims data of rehospitalization for any cause

CONTACTS AND LOCATIONS:
Overall Officials: Michael K Ong, MD, PhD, Principal Investigator — University of California, Los Angeles
Locations (6):
- United States (6):
  - University of California, Davis, Davis, California
  - University of California, Irvine, Irvine, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California
  - University of California, San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California

REFERENCES:
- [Background] Black JT, Romano PS, Sadeghi B, Auerbach AD, Ganiats TG, Greenfield S, Kaplan SH, Ong MK; BEAT-HF Research Group. A remote monitoring and telephone nurse coaching intervention to reduce readmissions among patients with heart failure: study protocol for the Better Effectiveness After Transition - Heart Failure (BEAT-HF) randomized controlled trial. Trials. 2014 Apr 13;15:124. doi: 10.1186/1745-6215-15-124. PMID 24725308
- [Derived] Ong MK, Romano PS, Edgington S, Aronow HU, Auerbach AD, Black JT, De Marco T, Escarce JJ, Evangelista LS, Hanna B, Ganiats TG, Greenberg BH, Greenfield S, Kaplan SH, Kimchi A, Liu H, Lombardo D, Mangione CM, Sadeghi B, Sadeghi B, Sarrafzadeh M, Tong K, Fonarow GC; Better Effectiveness After Transition-Heart Failure (BEAT-HF) Research Group. Effectiveness of Remote Patient Monitoring After Discharge of Hospitalized Patients With Heart Failure: The Better Effectiveness After Transition -- Heart Failure (BEAT-HF) Randomized Clinical Trial. JAMA Intern Med. 2016 Mar;176(3):310-8. doi: 10.1001/jamainternmed.2015.7712. PMID 26857383